CLINICAL TRIAL: NCT02348645
Title: Decompression Alone vs. Decompression and Instrumented Fusion for the Management of Lumbar Spinal Stenosis Associated With Stable Degenerative Spondylolisthesis: A Pragmatic Randomized Clinical Pilot Trial
Brief Title: Decompression vs. Fusion for Stable Degenerative Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-6927
Record Dates: First submitted 2014-09-09; First posted 2015-01-28 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Spinal Stenosis; Spondylolisthesis
Keywords: Pilot projects; Feasibility studies; Intervention studies; Orthopedics; Orthopedic Procedures; Neurosurgical Procedures; Neurosurgery; Spine; Spinal Fusion; Spondylodesis; Spondylosyndesis; Laminectomy; Foraminotomy; Decompression, surgical; Low Back Pain; Quality of Life
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Low Back Pain | interventions — Spinal Fusion; Laminectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decompression with fusion (Active Comparator): Spinal decompression surgery with instrumented spinal fusion
  Interventions: Procedure: Spinal fusion; Procedure: Spinal decompression
- Decompression alone (Active Comparator): Midline-sparing spinal decompression alone
  Interventions: Procedure: Spinal decompression

INTERVENTIONS:
Procedure: Spinal fusion
  Arms: Decompression with fusion
Procedure: Spinal decompression

SUMMARY:
The purpose of this study is to assess the feasibility of a full-scale multicenter randomized, controlled trial comparing the effectiveness of two surgical treatments for a condition associated with lumbar spinal stenosis called degenerative lumbar spondylolisthesis. Both treatments are currently used, but individual surgeons use different selection criteria for each treatment and use the procedures at different rates. The two procedures are decompression with fusion (the most common surgical procedure for spondylolisthesis) and midline-sparing decompression alone (which is also a standard treatment, but is not as widely used for treating spondylolisthesis). The investigators plan to collect the evidence on the following:

1. The feasibility of the trial protocol, and
2. Preliminary data on the effectiveness of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed to be surgical candidates with focal (1-2 level) lumbar spinal stenosis (LSS) and associated stable degenerative spondylolisthesis with the following characteristics:

  1. a clinical history of back, buttock and leg pain with walking or standing that is improved when lying, sitting or bending forward
  2. a clinical history of leg symptoms that are greater than or equal to back symptoms with walking or standing, and
  3. greater than 6 months of symptoms with failed conservative care
* aged 50 or over
* sufficient fluency in English or French to provide informed consent and complete questionnaires with or without the need of an interpreter

Exclusion Criteria:

* Greater than 25% listhesis or spinal instability as demonstrated by motion (>5mm of translation) on flexion extension radiographs or non-loaded (MRI/CT or supine x-rays) to loaded imaging (standing radiograph)
* Presence of kyphosis (>0 degrees at the affected level or globally), degenerative scoliosis (>10 degree using the Cobb method) with rotatory or lateral listhesis on preoperative x-rays
* Clinical history of osteoporotic fracture or chronic oral steroid use
* Previous posterior lumbar spinal surgery (excluding prior microdiscectomy)
* Patients who have evidence of neurological disorders that affect physical function (e.g. peripheral neuropathy), neuromuscular disorders (e.g. multiple sclerosis, Parkinson's etc.) or systemic illness (e.g. inflammatory arthritis) that affects physical function

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients recruited | 1 year
Number of eligible patients | 1 year
Reasons for refusal to consent | 1 year
Proportion of patients who adhere to randomized allocation | 2 years
Number of patients refusing to consent due to blinding | 1 year
Blinding status | 1.5 months post-surgery
  Patient's assessment of which treatment they received
Oswestry Disability Index (ODI) | 6-18 weeks, 6 months (optional), 12 months, and 24 months post-surgery
  10-item patient-reported questionnaire measuring disability related to low back pain. Each item has six response options ranging from 0 to 5; the responses are summed and rescaled so 0 indicates no disability and 100 indicates extreme disability.
Proportion of patients who receive randomized allocation | 2 years
Number of patients refusing to consent due to randomization | 1 year
Number, type and severity of adverse events | End of hospital stay (average 6.5 days post-surgery)

SECONDARY OUTCOMES:
Short-Form 12 scores: Physical Function, Bodily Pain, Physical Component Summary | Baseline; 6-18 weeks, 6 months (optional), 12 months, and 24 months post-surgery
  12-item patient-reported questionnaire for general health status based on the SF-36 Health Survey (version 2). Measures eight health domains, each scored so 0 is the worst and 100 is the best possible score: general health (GH), physical function (PF), bodily pain (BP), role limitations due to physical problems (RP), role limitations due to emotional problems (RE), mental health (MH), social functioning (SF), and energy/fatigue (VT). The domain scores can be aggregated into Physical Component Summary (PCS) and Mental Component Summary (MCS) scores, also scaled so 0 is the worst and 100 is the best possible score. This study will focus primarily on the Physical Function domain, the Bodily Pain domain, and the Physical Component Summary score.
Euro-QoL health utility index | Baseline; 6-18 weeks, 6 months (optional), 12 months, and 24 months post-surgery
  Patient-reported questionnaire for general health state which includes five items (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analog scale for self-rated health state. Using an existing U.S. population-based value set, responses will be converted to the corresponding health utility index (1.0=perfect health and 0.0=death).
Patient Health Questionnaire-9 score | Baseline
  Patient-reported questionnaire that measures severity of depression symptoms. It is scored from 0 to 27, with the following interpretation: 0-4=no symptoms, 5-9=minimal symptoms; 10-14=mild/minor depression or dysthymia; 15-19=moderate major depression; 20-27=severe major depression.
Costs incurred by patients | monthly from 1.5 to 12 months post-surgery; 24 months post-surgery
Hospital cost | End of hospital stay (average 6.5 days post-surgery)
Healthcare services used | Referral to 1 year post-surgery
  Other Ontario Health Insurance Plan (OHIP)-billed services used

CONTACTS AND LOCATIONS:
Overall Officials: Yoga Raja Rampersaud, MD FRCSC, Principal Investigator — University Health Network, Toronto; Anthony Perruccio, PhD, Principal Investigator — University Health Network, Toronto
Locations (8):
- Canada (8):
  - Foothills Medical Centre, Calgary, Alberta
  - Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec